CLINICAL TRIAL: NCT01972867
Title: A Pilot Study in Human Subjects Evaluating the Use of the NanoKnife System for Ablation of Prostate Cancer Tissue in an Intermediate Risk Patient Population
Brief Title: Study of NanoKnife for Ablation of Prostate Cancer in Intermediate Risk Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Angiodynamics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ON-NK310
Record Dates: First submitted 2013-10-23; First posted 2013-10-31 (Estimated); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Prostate Cancer
Keywords: Focal; Prostate; Cancer; Irreversible; Electroporation; NanoKnife
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- NanoKnife Procedure (Experimental): The NanoKnife procedure will be performed on focal prostate tumors, under ultrasound guidance.
  Interventions: Device: NanoKnife Procedure

INTERVENTIONS:
Device: NanoKnife Procedure — Subjects will be placed in the dorsal lithotomy position, under sterile technique. The NanoKnife procedure will be carried out under general anesthesia. A Foley catheter will be placed to aid in draining the bladder during treatment.
  Other Names: NanoKnife

SUMMARY:
The purpose of this study is to evaluate the feasibility and short-term safety and effectiveness of the NanoKnife System when used to ablate localized prostate cancer in intermediate risk subjects with organ-confined prostate cancer. This study will evaluate the feasibility of the NanoKnife System as a focal therapy.

DETAILED DESCRIPTION:
This study will involve six (6) subjects who meet the intermediate risk prostate cancer criteria defined by this protocol. The biopsy and imaging techniques that we will adopt within this trial are multiparametric MRI (mpMRI) and transperineal prostate biopsy (template mapping and/or limited targeted). The subjects' prostate cancer foci, the location of which will be determined by ultrasound guided transperineal prostate biopsy, will be targeted for treatment with the NanoKnife System. The primary objective of this the study will be to evaluate procedural and short-term post treatment safety of the NanoKnife treatment via incidence of adverse events and evaluation of effect on urologic (urinary and erectile) function. The secondary objective of this study is to evaluate the short term efficacy of the NanoKnife treatment. Local efficacy in the area of treatment will be assessed by histological evaluation of transperineal prostate biopsy cores at six (6) months post NanoKnife treatment, to evaluate the ablation zone created by the NanoKnife treatment. Other secondary outcomes include health-related quality of life levels evaluated using validated patient questionnaires. Following the 6 month transperineal prostate biopsy and mpMRI assessment, the data from these 6 subjects will be submitted to FDA for confirmation of short term safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Has at least a 10-year life expectancy
2. Have histologically confirmed organ-confined prostate cancer - clinical Stage ≤ T2c
3. Have a PSA ≤ 15 ng/mL or PSA density < 0.15 ng/mL2 if PSA is > 15 ng/mL
4. Has Gleason score 3+4 or 4+3
5. Has 10 mm or less of cancer-bearing prostate tissue in any biopsy core
6. No evidence of extraprostatic extension or seminal vesicle invasion by mpMRI
7. Able to visualize prostate gland adequately on transrectal ultrasound imaging during enrollment evaluation
8. Transperineal targeted prostate biopsies of lesion, plus 12 core systematic biopsies to include adequate sampling of the peripheral zone correlating with an intermediate risk lesion in the area of the MR-visible lesion.
9. A visible lesion on mpMRI that is accessible to Irreversible Electroporation (IRE) treatment
10. A non-MRI visible lesion detected via systematic standard biopsy will not be considered an exclusion condition provided the non-MRI visible lesion is singularly located in the contralateral hemisphere of the prostate; is Gleason 6; and comprises no more than 6mm linear extent of cancer-bearing tissue in a single core on standard biopsy.
11. Must sign a written informed consent
12. Understands and accepts the obligation and is logistically able to present for all scheduled follow-up visits

Exclusion Criteria:

1. Have known hypersensitivity to pancuronium bromide, atricurium or cisatricurium
2. Unfit for anesthesia or have a contraindication for agents listed for paralysis
3. Have an active urinary tract infection (UTI)
4. Have a history of bladder neck contracture
5. Are interested in future fertility
6. Have a history (within 3 years) of inflammatory bowel disease
7. Have a concurrent major debilitating illness
8. Had a malignancy within 5 years, including malignant melanoma, except for prostate cancer or other types of skin cancer
9. Have any active implanted electronic device (e.g., pacemaker)
10. Are unable to catheterize due to a urethral stricture disease
11. Have had prior or current prostate cancer therapies:

    1. Biologic therapy for prostate cancer
    2. Chemotherapy for prostate cancer
    3. Hormonal therapy for prostate cancer within three months of procedure
    4. Radiotherapy for prostate cancer
    5. Surgery for prostate cancer
12. Have had prior transurethral prostatectomy (TURP), stricture surgery, urethral stent or prostatic implants
13. Have had prior major rectal surgery (except hemorrhoids)
14. Unfit for pelvic MRI scanning (e.g., severe claustrophobia, permanent cardiac pacemaker, metallic implants that are likely to contribute significant image artifacts, allergy or contraindication to gadolinium (to enhance MRI)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-05-13 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Treatment procedural and short-term post-treatment safety profile | 6 months
  To determine the NanoKnife treatment procedural and short-term post-treatment safety profile by evaluating adverse event incidence, type, duration, severity and relationship to study device.
Treatment Morbidity Profile | 6 months
  To determine the NanoKnife treatment morbidity profile by evaluating urinary and erectile function.

SECONDARY OUTCOMES:
Completeness of Ablation | 6 months
  To determine completeness of ablation in the targeted prostate cancer tissue, in relation to probe placement and treatment parameters applied, as determined by histological evaluation of transperineal prostate biopsy cores at six (6) months post- treatment.
  * Determine post-treatment PSA kinetics
  * Determine effectiveness of therapy by post-treatment imaging (necrosis, presence of residual tissue)
  * Determine effectiveness of therapy by rates of biochemical and clinical progression; need for secondary or adjuvant treatment
Prostate-Specific Antigen Kinetics | 24 months
  Determine post-NanoKnife treatment prostate-specific antigen (PSA) kinetics including time to PSA nadir and post-nadir PSA stability.
Effectiveness of Therapy | 24 months
  To determine the effectiveness of therapy by post-treatment early-contrast MRI and multiparametric magnetic resonance imaging (mpMRI) to evaluate the area of necrosis and presence of residual tissue.
Effectiveness of Therapy | 24 months
  To determine the effectiveness of therapy by recording the rates of biochemical and clinical progression and the need for secondary or adjuvant treatment following therapy.
Health-Related Quality of Life | 24 months
  To determine health-related quality of life (HRQoL) levelsafter NanoKnife using validated patient questionnaires.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Rush University Medical Center, Chicago, Illinois
  - Mayo Clinic, Rochester, Minnesota